CLINICAL TRIAL: NCT07169604
Title: PERIOPERATIVE EFFECTS OF SPINAL ANALGESIA REGIMEN FOR ROBOTIC HYSTERECTOMY: A RETROSPECTIVE ANALYSIS
Brief Title: Analgesia Robotic Gynaecological Surgery
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Azienda Ospedaliero Universitaria, Santa Maria della Misericordia di Udine, Italy (Other)
Responsible Party: Principal Investigator, RUSSO ANDREA, medical doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3307
Record Dates: First submitted 2025-08-19; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
we will retrospectively investigate the effect of intratecal morphine administration on postoperative pain relief for patients scheduled for robotic hysterectomy

ELIGIBILITY:
Inclusion Criteria:

patients scheduled for robotic hysterectomy acceptation of written informed consent

Exclusion Criteria:

were contraindications to neuraxial anesthesia (such as coagulopathies, platelet count below 100,000/mm³ or thrombocytopathy), severe valvular heart disease, left ventricular ejection fraction less than 35%, history of obstructive or restrictive pulmonary disease, or significant neurological disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: patients with gynaecological malignant or benign condition needed for hysterectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
pain scores | admission at PACU admission, discharge from PACU, 24 hours after surgery (T2)
  we will registered the visual analogue scale number

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Policlinico Gemelli, Roma, RM, Italy